CLINICAL TRIAL: NCT03475238
Title: Nursing Research on the Occurrence of Serious Adverse Events in Intensive Care Unit During Bed Bath and Nursing Care. NURSIE Study
Brief Title: Analysis of Factors Related to Occurrence of Serious Adverse Events During Nursing in Intensive Care Units
Acronym: NURSIE
Status: Completed | Type: Observational
Sponsor: French Society for Intensive Care (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-A00046-49
Record Dates: First submitted 2018-03-11; First posted 2018-03-23 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Nursing Caries; Critical Care
Keywords: critical care
MeSH Terms: interventions — Nursing Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort for nursing care: Patients in ICU under oxygen and/or mechanical ventilation and/or vasoactive drugs and/or non-invasive ventilation
  Interventions: Procedure: Nursing care

INTERVENTIONS:
Procedure: Nursing care — The nursing care will be defined as a lateral mobibization and a length of care superior or equal to 10 min

SUMMARY:
Patients who are hospitalized in intensive care unit (ICU) require basic nursing care to improve patient hygiene, to promote comfort, to prevent pressure ulcer, and foot or hand's retractations.

Those nursing cares require mobilization very frequently which expose critically ill patients to occurrence of serious adverse events (SAE) such as i) hemodynamic, neurologic, and respiratory variations ii) unplanned dislodgement (lines, drains, catheters, endotracheal tube..)

Few study have evaluated relation between SAE occurence and several patient's, service's, health-care provider's caracteristics. We plan to analyse those factors to find some ways to prevent SAE occurence during nursing and hygiene cares.

ELIGIBILITY:
Inclusion Criteria:

* Health-care affiliated
* Length of ICU stay < 72 h
* Patient with endotracheal tube
* Patient with tracheostomy
* Patient receiving vasoactives drugs (norepinephrine, epinephrine, Dobutamine)
* Patient undergoing no invasive ventilation during 1hour minimum of 24 hours before the selection
* Patient undergoing hight flow oxygen therapy heated and humidified

Exclusion Criteria:

* Patient already included in this study
* Medical contraindication to the bed bath with lateral mobilization
* Withdrawal of life sustaining treatment
* Spinal trauma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Each participating unit will include all consecutive patients staying in the ICU.
  Each day a screening of the patients will be released between 8 and 10 am.
Sampling Method: Probability Sample
Enrollment: 262 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2018-07-15 (Actual); Study Completion 2019-02-13 (Actual)

PRIMARY OUTCOMES:
Incidence of occurrence of at least one serious avderse event (SAE) (defined below) during the nursing care while the study period (72 hours) | 72 hours
  Determinate incidence of occurrence of at least one SAE (defined below) during the nursing care while the study period (72 hours) The nursing care will be defined as a lateral mobibization and a length of care sup or equal to 10min
  SAE are considered according to litterature as :
  * Cardiac arest
  * Unplanned extubation
  * Episode of Spo2 riequiring therapeutic intervention
  * Artificial airway obstruction requiring endotracheal suctionning
  * Unplanned dislodgements related to lines or catheters drains
  * Hypotension with therapeutic intervention
  * Cardiac rhythm disorders with therapeutic intervention
  * Agitation with therapeutic intervention
  * Equipment failure or dysfunction
  * Patient fall
  * Need for doctor help
  * Increased intracranial pressure > 20 mmHg
  * Acute painful crisis

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu Lloung, Study Director — French Intensive Care Society; Jean Baptiste Lascarrou, MD, Study Chair — French Intensive Care Society
Locations (26):
- Belgium (3):
  - Hopital de Bruxelles, Brussels
  - CHU Charleroi, Charleroi
  - Hopital Civil Marie Curie, Charleroi
- France (21):
  - CH Andre Migniot, Versailles, A
  - CHU Besançon, Besançon
  - CHU Ambroise Paré, Boulogne-Billancourt
  - CH Sud Francilien, Corbeil-Essonnes
  - CH de Dax, Dax
  - CH de la Dracénie, Draguignan
  - CHRU Lille, Lille
  - Hopital Jeanne De Flandre, Lille
  - CHU Marseille, Marseille
  - CHU Nantes, Nantes
  - CHU Nice, Nice
  - CHU Nimes, Nîmes
  - CHR Orléans, Orléans
  - CHU La Pitié Salpétrière, Paris
  - CHU Lariboisière, Paris
  - CHU Necker Enfant Malade, Paris
  - Hopital Europeen George Pompidou, Paris
  - CHU Strasbourg, Strasbourg
  - CHU Toulouse, Toulouse
  - CH Valence, Valence
  - CHI Lucie & Raymond Aubrac, Villeneuve-Saint-Georges
- Centre Hospitalier Emile Mayrisch, Luxembourg, Luxembourg
- Hopital de la Tour, Meyrin, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided